CLINICAL TRIAL: NCT03855865
Title: A Randomized, Double-blind, Placebo- and Active- Controlled, Multicenter Study of Rapastinel as Monotherapy in Major Depressive Disorder
Brief Title: Study of Rapastinel as Monotherapy in Major Depressive Disorder (MDD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-MD-31; 2018-000063-88 (EudraCT Number)
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide; Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel (Experimental): Rapastinel (450 mg prefilled syringe, weekly intravenous IV administration).
  Interventions: Drug: Rapastinel
- Vortioxetine (Active Comparator): Vortixetine (10 mg with available dose increase to vortioxetine 20 mg oral daily after 3 weeks of administration).
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Placebo (prefilled syringe, weekly IV administration or oral daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel (prefilled syringe, weekly intravenous IV administration).
  Arms: Rapastinel
Drug: Vortioxetine — Vortixetine (10 mg with available dose increase to vortioxetine 20 mg oral daily after 3 weeks of administration).
  Arms: Vortioxetine
Drug: Placebo — Placebo (prefilled syringe, weekly IV administration or oral daily).
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy, safety, and tolerability of 450 milligrams (mg) of Rapastinel, compared to 10 mg of Vortixetine and placebo in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1
* Have inadequate response to 1-3 antidepressant therapies given at adequate dose and duration in the current episode
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:

  1. Schizophrenia spectrum or other psychotic disorder
  2. Bipolar or related disorder
  3. Major neurocognitive disorder
  4. Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
  5. Dissociative disorder
  6. Posttraumatic stress disorder
  7. MDD with psychotic features
* Significant suicide risk, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at the End of the Double Blind Treatment Period (DBTP) (end of Week 6) | Baseline to end of Week 6
  The MADRS, a clinician-rated scale, will be used to assess depressive symptomatology. Participants are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item will be scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity.

SECONDARY OUTCOMES:
Change from Baseline in MADRS Total Score at Day 1 Post-first Dose of Treatment | Baseline to Day 1 post-first dose
  The MADRS, a clinician-rated scale, will be used to assess depressive symptomatology. Participants are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item will be scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Debelle, Study Director — Allergan

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://AllerganClinicalTrials.com